CLINICAL TRIAL: NCT03527758
Title: Correlation Between Circulating Biomarkers of Organs Damage and Intraoperative Hypotension Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Catania (Other)
Collaborators: Giovanni Li Volti (Unknown); Marinella Astuto (Unknown); Francesco Vasile (Unknown); Gaetano Joseph Palumbo (Unknown); Mirko Mineri (Unknown); Christian Bonsignore (Unknown); Salvatore Pennisi (Unknown); Carmelo Minardi (Unknown); Bruno Lanzafame (Unknown); Luigi Lavia (Unknown); Veronica Dezio (Unknown)
Responsible Party: Principal Investigator, Paolo Murabito, Assistant Professor, University of Catania
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 46/2018/PO
Record Dates: First submitted 2018-04-27; First posted 2018-05-17 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Hypotension; Brain Injuries; Renal Failure; Endothelial Dysfunction
Keywords: Biomarkers; Hypotension; Organ Protection; Intraoperative
MeSH Terms: conditions — Hypotension; Brain Injuries; Renal Insufficiency

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Invasive intraoperative monitoring (No Intervention)
- Flo TracIQ with HPI software (Experimental)
  Interventions: Device: Flo TracIQ with HPI software

INTERVENTIONS:
Device: Flo TracIQ with HPI software — Patients will be monitored intraoperatively with Flo TracIQ with HPI software in order to predict hypotensive events. Blood sample will be obtained in order to evaluate ealy organ dysfunction.
  Arms: Flo TracIQ with HPI software

SUMMARY:
Intraoperative hypotension (defined as mean arterial pressure below 65 mmHg) is associated with increased organs dysfunction and mortality. Even short durations of reduced arterial blood pressure episodes significantly increased the risk of myocardial injury, neurological deficits, renal failure, and mortality. Hypotension rate during surgery is quite common and recent studies showed an incidence up to 60% of patients endured hypotension during anesthesia for an average of 10% of surgical time.

Nowadays hypotension seems to be preventable even if current management of the hypotensive episodes is predominantly reactive and rather occurs with some delay.

The investigators hypothesize that the prevention of hypotension by means Edwards Lifesciences new technology (HPI software) can improve patients outcome after surgery.

The present pilot randomized clinical trial is aimed at investigating various biomarkers involved in organ dysfunction and how they correlate with different intraoperative hypotension management strategies (Invasive blood pressure monitored by a normal arterial line vs Invasive blood pressure monitored by Edwards FloTracIQ system with HPI software).

DETAILED DESCRIPTION:
The primary objective of this pilot study is to investigate if an early treatment of intraoperative hypotension driven by an Edwards Lifesciences new technology (Hypotension Probability Index - HPI software) and integrated hemodynamic variables is able to determine a modification of the blood levels of several specific biomarkers of tissue and organ damage compared to a traditional management of hypotension. It will also be evaluated if the management strategy of patient hemodynamics based on the Hypotension Probability Index (HPI) is associated with a lower incidence of hypotensive events and / or a shorter overall duration of intraoperative hypotension.

In the study will be enrolled forty adult patients requiring an arterial line (at discretion of treating physician) undergoing non-cardiac non-day surgery (with an expected duration of more than 2 hours and an aimed medium arterial pressure - MAP of 65 mmHg) at the Universitary Hospital of Catania.

The patients will be randomly (1:1) assigned to one of the subsequent two groups: a group monitored with FloTracIQ with HPI software (Treatment Group) and a group with standard invasive blood pressure monitoring (Control Group).

In the Control Group, all hypotensive episodes during surgery will be treated according to standard of care.

Patients randomized to the Treatment Group will receive monitoring with integration of HPI index and hemodynamic parameters visible on the EV1000 platform; these informations will be used to guide the investigator in the choice of the more appropriate treatment to be carried out. The value of HPI is updated every 20 seconds and expresses in percentage the probability of occurrence of a hypotensive event. The cut-off value of HPI is equal to 85%. Values above the cut-off are related to a higher probability of hypotension. A specific visual and sound "ALERT" will indicate to the investigator if the threshold value is reached / exceeded. Any treatment strategy will be based on integrated analysis of clinical and instrumental data showed on the screen of the EV1000 platform [MAP, cardiac output (CO), systemic vascular resistance (SVR), stroke volume (SV), stroke volume variation (SVV), intra-ventricular pressure rate of rise (dP/dt), dynamic arterial elastance (Eadyn)].

In both groups different blood samplings will be performed in order to assess biomarkers of specific organ dysfunction: T0 (baseline, before starting operating procedures); T1 (2 hours after starting anesthesia); T2 (at the end of surgical procedures). The following biomarkers will be assessed: neuron specific enolase and S100B (for brain monitoring); high sensitive cardiac troponin T (for heart monitoring); Neutrophil Gelatinase-Associated Lipocalin (NGAL, for kidney monitoring); circulating endothelial cells counting and cytofluorimetric analysis (for endothelial monitoring). There will also be determined the systemic effect of intraoperative hypotension as measured by inflammatory cytokines [Interleukin (IL)-6, IL-1 beta and Tumor necrosis factor (TNF)-alfa], oxidative stress (reduced glutathione, lipid hydroperoxides) and markers of hypoxia (HIF1alpha, lactate, acetylCoA, CoA).

Various clinical informations will be collected at the same time: glomerular filtration rate, plasma electrolytes, creatinine, aspartate aminotransferase (AST), alanine aminotransferase (ALT), blood gasses analysis, anion gap.

A telephone interview will be performed one month after surgery, in order to investigate general health condition and any re-admission to hospital.

Sample size calculation:

Given the pilot nature of the study, no formal justification of sample size has been made.

Statistical analysis:

For a test of normal distribution, the Kolmogorov-Smirnov test will be used. Continuous data with normal distribution will be tested with paired or unpaired t tests, non-normally distributed data using Mann-Whitney U test and Wilcoxon rank-sum test for unpaired and paired results, respectively.

Changes in biomarkers over time will be tested using analysis of variance (ANOVA) on repeated measurements. Categorical data will be tested using Chi-square test and Chi-square test for trend. Data will be presented as mean ± standard deviation when normally distributed and as median [interquartile ranges] in case of abnormal distribution. A p < 0.05 will be considered statistically significant for all tests.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older;
* Planned for elective non-cardiac non-day surgery with an expected duration of more than 2 hours;
* Planned to receive general anesthesia;
* Planned to receive an arterial line during surgery;
* Aim for MAP of 65 mmHg during surgery;
* Being able to give written informed consent prior to surgery.

Exclusion Criteria:

Age less than 18 years;

* Aim for MAP other than 65 mmHg at discretion treating physician;
* Significant hypotension before surgery defined as a MAP <65;
* Right- or left sided cardiac failure [e.g. left ventricular ejection fraction (LVEF)<35%];
* Known cardiac shunts (significant);
* Known aortic stenosis (severe);
* Severe cardiac arrhythmias including atrial fibrillation;
* Chronic kidney disease (as chronic kidney disease may affect the interpretation and prognostic significance of changes in urinary biomarkers);
* Liver surgery;
* Vascular surgery with clamping of the aorta;
* Diabetes.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2020-01-15 (Actual)

PRIMARY OUTCOMES:
Variation from basal of the levels of biomarkers of brain, heart, kidney and endothelial injury. | 2 hours after starting anesthesia
  The following biomarkers will be assessed: neuron specific enolase and S100B (for brain monitoring); high sensitive cardiac troponin T (for heart monitoring); Neutrophil Gelatinase-Associated Lipocalin (NGAL, for kidney monitoring); circulating endothelial cells counting and cytofluorimetric analysis (for endothelial monitoring).Systemic effects of intraoperative hypotension will be determine by measuring inflammatory cytokines (IL-6, IL-1 beta and TNF-alfa), oxidative stress biomarkers (reduced glutathione, lipid hydroperoxides) and markers of hypoxia (HIF1alpha, lactate, acetylCoA, CoA).
Variation from basal of the levels of biomarkers of brain, heart, kidney and endothelial injury. | End of surgical procedures
  The following biomarkers will be assessed: neuron specific enolase and S100B (for brain monitoring); high sensitive cardiac troponin T (for heart monitoring); Neutrophil Gelatinase-Associated Lipocalin (NGAL, for kidney monitoring); circulating endothelial cells counting and cytofluorimetric analysis (for endothelial monitoring).Systemic effects of intraoperative hypotension will be determine by measuring inflammatory cytokines (IL-6, IL-1 beta and TNF-alfa), oxidative stress biomarkers (reduced glutathione, lipid hydroperoxides) and markers of hypoxia (HIF1alpha, lactate, acetylCoA, CoA).

SECONDARY OUTCOMES:
Incidence of hypotension during surgery | End of surgical procedures
Time spent in hypotension during surgery | End of surgical procedures
Patient-reported outcomes | 30 days postsurgical procedure
  A telephone interview will be performed in order to investigate general health conditions and any re-admission to hospital.

CONTACTS AND LOCATIONS:
Locations (1):
- "G. Rodolico" Presidium of the Azienda Ospedaliero Universitaria "Policlinico-Vittorio Emanuele", Catania, Italy

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR